CLINICAL TRIAL: NCT01537601
Title: Effect of Circumcision on the Risk of Febrile Urinary Tract Infections in Children With Posterior Urethral Valves.
Brief Title: CIRCumcision and Urinary Tract Infections in Boys With Posterior Urethral Valves
Acronym: CIRCUP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012/CHR/01
Record Dates: First submitted 2012-02-17; First posted 2012-02-23 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Posterior Urethral Valves
Keywords: Posterior urethral valves; Febrile urinary tract infection; Circumcision; Antibioprophylaxis; Impact on family
MeSH Terms: interventions — Circumcision, Male; Antibiotic Prophylaxis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antibiotic prophylaxis alone (Other): Children will be on antibioprophylaxis and will not have a circumcision.
  Interventions: Other: Antibiotic prophylaxis alone
- Circumcision and antibiotic prophylaxis (Experimental): Children will have a circumcision at the time of valve resection and will be on antibioprophylaxis
  Interventions: Procedure: Circumcision

INTERVENTIONS:
Procedure: Circumcision — Circumcision
  Arms: Circumcision and antibiotic prophylaxis
Other: Antibiotic prophylaxis alone — Antibiotic prophylaxis alone
  Arms: Antibiotic prophylaxis alone

SUMMARY:
Children with posterior urethral valves (PUV) are at risk of presenting febrile urinary tract infections (UTI). Circumcision has been shown to decrease the number of febrile UTIs in healthy children. The effect of circumcision on the number of UTIs in boys with PUV has not yet been studied. Through a prospective randomised trial of children with posterior urethral valves the investigators wish to determine the effect of circumcision on the risk of presenting febrile UTIs. One group will be on antibiotic prophylaxis alone and the other will be on antibiotic prophylaxis plus circumcision performed at the time of valve resection. Both groups will be followed for two years, with clinical examination at 1, 3, 6, 12, 18 and 24 months. A DMSA scan will be performed at 1-2 and 24 months and biological renal function will also be monitored. The relative risk of presenting a febrile UTI in each group will be determined. Clinical, radiological and antenatal data concerning each child will be analysed. At 24 months follow-up, an "impact on family scale" survey (IOFS) will be proposed parents.

DETAILED DESCRIPTION:
After diagnosis of posterior urethral valves, children will be randomised either to antibioprophylaxis alone or antibioprophylaxis plus circumcision. Circumcision will be performed at the time of valve resection. Children will undergo a cystogram between 1 and 4 months to control valve resection. They will be followed for two years and the number of febrile UTIs in each group will be compared. The diagnosis of febrile UTI will be confirmed by urethral catheterisation or suprapubic aspiration. A DMSA scan will be performed at the beginning and end of the study to determine whether children who have presented febrile UTIs show deterioration of their DMSA as compared to those who did not present febrile UTIs.

At 24 months follow-up, "impact on family scale" survey (IOFS) whose main objective is to evaluate the impact of family support for a child with posterior urethral valves will be proposed parents.

ELIGIBILITY:
Inclusion Criteria:

* male
* aged 0 to 28 days
* diagnosed with posterior urethral valves within the 28 first day of life
* holders of parental authority affiliated to French national health insurance
* informed consent signed by holders of parental authority

Exclusion Criteria:

* boys with hypospadias or epispadias or any other anomaly rendering circumcision impossible
* concomitant participation to another clinical trial

Max Age: 28 Days | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02-18 (Actual)

PRIMARY OUTCOMES:
Relative risk of presenting a febrile UTI | 24 months

SECONDARY OUTCOMES:
Number of children with febrile UTIs in each group at two years | 24 months
Evolution of compliance to antibioprophylaxis. | 24 months
Evolution of the grade of reflux | At diagnosis and at 3 months
Comparison of the number of children who will show deterioration of their DMSA scan between children who have had UTIs and those who have not. | 24 months
number and type of adverse effects related to circumcision and antibiotic prophylaxis | 24 months
Identification of the responsible bacteria | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Frédérique Sauvat, MD, Principal Investigator — Regional Hospital Reunion Island - Felix Guyon Site; Eric Dobremez, MD, Principal Investigator — CHU Bordeaux, Hôpital Pellegrin Enfants; Laurent Fourcade, MD, Principal Investigator — CHU Limoges - Hôpital de la mère et de l'enfant; Nicolas Kalfa, MD, Principal Investigator — CHU Montpellier - Hôpital Lapeyronie; Frédéric Auber, MD, Principal Investigator — CHU St Jacques - Besançon; Benjamin Frémond, Principal Investigator — CHU Rennes; Alaa El Ghoneimi, MD, Principal Investigator — CHU Robert Debré; Thomas Blanc, MD, Principal Investigator — CHU de Necker Enfants Malades; Jean Michel Guys, MD, Principal Investigator — Hôpital d'enfants de la Timone, Marseille; Thierry Merrot, MD, Principal Investigator — CHU Nord, Marseille; Marc David Leclair, MD, Principal Investigator — Nantes University Hospital; Georges Audry, MD, Principal Investigator — CHU Armand Trousseau, Paris; Marie-Laurence Poli-merol, MD, Principal Investigator — CHU de Reims
Locations (1):
- Department of pediatric surgery, Bordeaux hospital, Bordeaux, France

REFERENCES:
- [Background] Woolf AS, Thiruchelvam N. Congenital obstructive uropathy: its origin and contribution to end-stage renal disease in children. Adv Ren Replace Ther. 2001 Jul;8(3):157-63. doi: 10.1053/jarr.2001.26348. PMID 11533916
- [Background] Parkhouse HF, Barratt TM, Dillon MJ, Duffy PG, Fay J, Ransley PG, Woodhouse CR, Williams DI. Long-term outcome of boys with posterior urethral valves. Br J Urol. 1988 Jul;62(1):59-62. doi: 10.1111/j.1464-410x.1988.tb04267.x. PMID 3408870
- [Background] Singh-Grewal D, Macdessi J, Craig J. Circumcision for the prevention of urinary tract infection in boys: a systematic review of randomised trials and observational studies. Arch Dis Child. 2005 Aug;90(8):853-8. doi: 10.1136/adc.2004.049353. Epub 2005 May 12. PMID 15890696
- [Background] Simforoosh N, Tabibi A, Khalili SA, Soltani MH, Afjehi A, Aalami F, Bodoohi H. Neonatal circumcision reduces the incidence of asymptomatic urinary tract infection: a large prospective study with long-term follow up using Plastibell. J Pediatr Urol. 2012 Jun;8(3):320-3. doi: 10.1016/j.jpurol.2010.10.008. Epub 2010 Nov 5. PMID 21115400
- [Background] Mukherjee S, Joshi A, Carroll D, Chandran H, Parashar K, McCarthy L. What is the effect of circumcision on risk of urinary tract infection in boys with posterior urethral valves? J Pediatr Surg. 2009 Feb;44(2):417-21. doi: 10.1016/j.jpedsurg.2008.10.102. PMID 19231547
- [Result] Harper L, Blanc T, Peycelon M, Michel JL, Leclair MD, Garnier S, Flaum V, Arnaud AP, Merrot T, Dobremez E, Faure A, Fourcade L, Poli-Merol ML, Chaussy Y, Dunand O, Collin F, Huiart L, Ferdynus C, Sauvat F. Circumcision and Risk of Febrile Urinary Tract Infection in Boys with Posterior Urethral Valves: Result of the CIRCUP Randomized Trial. Eur Urol. 2022 Jan;81(1):64-72. doi: 10.1016/j.eururo.2021.08.024. Epub 2021 Sep 22. PMID 34563412